CLINICAL TRIAL: NCT01205581
Title: Immunogenicity of Fluzone HD,A High Dose Influenza Vaccine, In Children With Cancer or HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLUHD
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-07

CONDITIONS: HIV; Cancer
Keywords: Fluzone; Trivalent Influenza Vaccine
MeSH Terms: conditions — Neoplasms; Influenza, Human | interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Leukemia-HD (Active Comparator): Subjects with a diagnosis of leukemia will be vaccinated twice with Fluzone High Dose Vaccine and evaluated for development of immune responses.
  Interventions: Biological: Fluzone High Dose Vaccine
- Leukemia-SD (Active Comparator): Subjects with a diagnosis of leukemia will be vaccinated twice with Fluzone Standard Dose Vaccine and evaluated for development of immune responses.
  Interventions: Biological: Fluzone Standard Dose Vaccine
- Solid Tumor-HD (Active Comparator): Subjects with a diagnosis of solid tumor will be vaccinated twice with Fluzone High Dose Vaccine and evaluated for development of immune responses.
  Interventions: Biological: Fluzone High Dose Vaccine
- Solid Tumor-SD (Active Comparator): Subjects with a diagnosis of solid tumor will be vaccinated twice with Fluzone Standard Dose Vaccine and evaluated for development of immune responses.
  Interventions: Biological: Fluzone Standard Dose Vaccine
- HIV-HD (Active Comparator): Subjects with a diagnosis of human immunodeficiency virus (HIV) will be vaccinated twice with Fluzone High Dose Vaccine and evaluated for development of immune responses.
  Interventions: Biological: Fluzone High Dose Vaccine
- HIV-SD (Active Comparator): Subjects with a diagnosis of human immunodeficiency virus (HIV) will be vaccinated twice with Fluzone Standard Dose Vaccine and evaluated for development of immune responses.
  Interventions: Biological: Fluzone Standard Dose Vaccine

INTERVENTIONS:
Biological: Fluzone High Dose Vaccine — Two doses of Fluzone HD will be administered to children with leukemia, solid tumor, or HIV.
  Other Names: Fluzone-HD
  Arms: HIV-HD; Leukemia-HD; Solid Tumor-HD
Biological: Fluzone Standard Dose Vaccine — Two doses of Fluzone Standard Dose Vaccine will be administered to children with leukemia, solid tumor, or HIV.
  Other Names: Fluzone-SD
  Arms: HIV-SD; Leukemia-SD; Solid Tumor-SD

SUMMARY:
This is an open label-study of Fluzone HD, a high-dose form of trivalent, inactivated influenza vaccine (TIV), vs. Fluzone, a standard-dose form of TIV. Subjects with cancer or HIV will be vaccinated twice with one of the two vaccines and evaluated for development of immune responses.

DETAILED DESCRIPTION:
The primary objectives of this study are to compare the immune response of Fluzone HD, a high-dose, trivalent influenza vaccine (TIV), to Fluzone, a standard-dose TIV, in children with cancer and in children with HIV.

The secondary objectives of this study are to:

* Describe the safety and reactogenicity of high-dose and standard-dose TIV.
* Compare the immunogenicity induced by 1 dose, compared to 2 doses, of high-dose and standard-dose TIV.
* Describe the relationship between baseline lymphocyte numbers/function and robustness/durability of the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 years (on or past their 3rd birthday) through 21 years of age (not yet reached their 22nd birthday) at the time of entry into the study.
* Written informed consent (and assent, if applicable) obtained.
* Participant has a diagnosis of cancer or HIV.
* If subject has cancer, currently receiving chemotherapy and /or radiotherapy for the treatment of cancer or has received chemotherapy in the past 12 weeks

Exclusion Criteria

* Severe hypersensitivity to egg proteins or any component of Fluzone, or life-threatening reactions after any previous administration of any influenza vaccine;
* History of Guillain-Barre´ syndrome in the subject or subject's family (parents, siblings, half siblings, or children);
* Not willing to agree to acceptable birth control for three months after study immunization

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A McCullers, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were ≥3-21 yrs. at study entry with diagnosis of cancer or HIV. Those with cancer were receiving chemotherapy and/or radiotherapy or had received chemotherapy in the prior 12 weeks. One participant was enrolled but was lost to follow up prior to randomization. 84 participants were randomized between 9/2010 and 10/2011.
Pre-assignment Details: Participants excluded if they had: pre-vaccination titer of ≥1:2560, severe hypersensitivity to egg proteins or any component of Fluzone, life-threatening reaction after prior influenza vaccine, history of Guillain-Barre syndrome in subject/subject's family, or unwilling to agree to acceptable birth control for 3 months after each dose.
Groups:
- Leukemia-HD: Patients with a diagnosis of leukemia who received the high dose Fluzone HD.
- Leukemia-SD: Patients with a diagnosis of leukemia who received the standard dose Fluzone.
- Solid Tumor-HD: Patients with a diagnosis of solid tumor who received the high dose Fluzone HD.
- Solid Tumor-SD: Patients with a diagnosis of solid tumor who received the standard dose Fluzone.
- HIV-HD: Patients with a diagnosis of HIV who received the high dose Fluzone HD.
- HIV-SD: Patients with a diagnosis of HIV who received the standard dose Fluzone.
Period: Overall Study
Arm/Group | Leukemia-HD | Leukemia-SD | Solid Tumor-HD | Solid Tumor-SD | HIV-HD | HIV-SD
Started | 14 | 13 | 8 | 9 | 20 | 20
Completed | 13 | 13 | 8 | 9 | 20 | 20
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was an open-label study where participants were randomized at a 1:1 ratio into Fluzone high-dose (HD) and Fluzone standard dose (SD) groups by disease group with the use of a computer-generated randomization schedule.
Groups:
- Total: Total of all reporting groups
Arm/Group | Leukemia-HD | Leukemia-SD | Solid Tumor-HD | Solid Tumor-SD | HIV-HD | HIV-SD | Total
Number analyzed (Participants) | 13 | 13 | 8 | 9 | 20 | 20 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (5.7) | 11.8 (5.1) | 12.4 (4.2) | 11.7 (4.5) | 16.7 (5.6) | 19.9 (1.8) | 14.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 4 | 7 | 4 | 28
  Male | 9 | 8 | 4 | 5 | 13 | 16 | 55

OUTCOME MEASURES:

1. Primary Outcome: Rate of Seroconversion After 1 Dose of Vaccine
Description: The immune response of Fluzone HD to Fluzone was determined using the hemagglutination-inhibition (HAI) assay to each of the 3 antigens contained in the vaccine: H1, H3 and B. Seroconversion was defined as a post-vaccine HAI titer ≥40 if baseline was <10, or a 4-fold rise in HAI titer if the baseline ≥10.
Time Frame: at least 21 days after first dose, which is given at the time of baseline evaluation visit, and prior to second dose
Population: Two patients in the HIV-HD group were excluded because data was only available at baseline. These 2 patients were lost for follow-up before evaluation for post-vaccine immune response.
Measure: Number; unit: percentage of participants
Arm/Group | Leukemia-HD | Leukemia-SD | Solid Tumor-HD | Solid Tumor-SD | HIV-HD | HIV-SD
Number analyzed (Participants) | 13 | 13 | 8 | 9 | 18 | 20
percentage of participants
  H1 antigen | 31 | 0 | 50 | 22 | 61 | 65
  H3 antigen | 77 | 85 | 50 | 89 | 72 | 65
  B antigen | 38 | 46 | 63 | 44 | 67 | 35

2. Secondary Outcome: Number of Participants Reporting Grade 3 and Grade 4 Adverse Events Possibly, Probably, or Definitely Attributable to Fluzone or Fluzone HD
Description: Number of participants reporting grade 3 and grade 4 adverse events possibly, probably, or definitely attributable to Fluzone or Fluzone HD.
Time Frame: From initial vaccine administration through up to 8 months
Population: Adverse events of Fluzone HD and Fluzone are provided as combined data from cancer and HIV patients, since there is no reason to believe one group is more susceptible to adverse events than the other.
Measure: Number; unit: participants
Groups:
- High-dose FluzoneHD: 41 participants received 80 doses of high-dose FluzoneHD.
- Standard Dose Fluzone: 42 participants received 82 doses of standard-dose Fluzone.
Arm/Group | High-dose FluzoneHD | Standard Dose Fluzone
Number analyzed (Participants) | 41 | 42
participants | 1 | 0

3. Secondary Outcome: Rate of Sero-conversion for 1 Dose vs. 2 Doses of Fluzone HD
Description: The rate of seroconversion to the 3 antigens contained in the vaccine was determined by hemagglutination-inhibition test and was compared by disease.
  The immune response of 1 dose vs. 2 doses of Fluzone HD was determined using the hemagglutination-inhibition (HAI) assay to each of the 3 antigens contained in the vaccine: H1, H3 and B. Seroconversion was defined as a post-vaccine HAI titer ≥40 if baseline was <10, or a 4-fold rise in HAI titer if the baseline ≥10.
Time Frame: at least 21 days after each dose of vaccine
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Leukemia-1 Dose: Patients with a diagnosis of leukemia who received one dose of high dose Fluzone HD.
- Leukemia-2 Doses: Patients with a diagnosis of leukemia who received 2 doses of high dose Fluzone HD.
- Solid Tumor-1 Dose: Patients with a diagnosis of solid tumor who received one dose of high dose Fluzone HD.
- Solid Tumor-2 Doses: Patients with a diagnosis of solid tumor who received 2 doses of high dose Fluzone HD.
- HIV-1 Dose: Patients with a diagnosis of HIV who received one dose of high dose Fluzone HD.
- HIV-2 Doses: Patients with a diagnosis of HIV who received 2 doses of high dose Fluzone HD.
Arm/Group | Leukemia-1 Dose | Leukemia-2 Doses | Solid Tumor-1 Dose | Solid Tumor-2 Doses | HIV-1 Dose | HIV-2 Doses
Number analyzed (Participants) | 13 | 13 | 8 | 8 | 18 | 18
percentage of participants
  H1 antigen | 31 | 54 | 50 | 88 | 61 | 72
  H3 antigen | 77 | 85 | 50 | 63 | 72 | 72
  B antigen | 38 | 85 | 63 | 75 | 67 | 78

4. Secondary Outcome: Rate of Sero-conversion for 1 Dose vs. 2 Doses of Fluzone SD
Description: The rate of seroconversion to the 3 antigens contained in the vaccine was determined by hemagglutination-inhibition test and was compared by disease.
  The immune response of 1 dose vs. 2 doses of Fluzone SD was determined using the hemagglutination-inhibition (HAI) assay to each of the 3 antigens contained in the vaccine: H1, H3 and B. Seroconversion was defined as a post-vaccine HAI titer ≥40 if baseline was <10, or a 4-fold rise in HAI titer if the baseline ≥10.
Time Frame: at least 21 days after each dose of vaccine
Measure: Number; unit: percentrage of participants
Groups:
- Leukemia-1 Dose: Patients with a diagnosis of leukemia who received one dose of high dose Fluzone SD.
- Leukemia-2 Doses: Patients with a diagnosis of leukemia who received 2 doses of high dose Fluzone SD.
- Solid Tumor-1 Dose: Patients with a diagnosis of solid tumor who received one dose of high dose Fluzone SD.
- Solid Tumor-2 Doses: Patients with a diagnosis of solid tumor who received 2 doses of high dose Fluzone SD.
- HIV-1 Dose: Patients with a diagnosis of HIV who received one dose of high dose Fluzone SD.
- HIV-2 Doses: Patients with a diagnosis of HIV who received 2 doses of high dose Fluzone SD.
Arm/Group | Leukemia-1 Dose | Leukemia-2 Doses | Solid Tumor-1 Dose | Solid Tumor-2 Doses | HIV-1 Dose | HIV-2 Doses
Number analyzed (Participants) | 13 | 13 | 9 | 9 | 20 | 20
percentrage of participants
  H1 antigen | 0 | 54 | 22 | 67 | 65 | 70
  H3 antigen | 85 | 92 | 89 | 89 | 65 | 70
  B antigen | 46 | 85 | 44 | 89 | 35 | 75

5. Secondary Outcome: Rate of Vaccine Response by Seroconversion Compared by Absolute Lymphocyte Count (ALC)
Description: The relationship between baseline lymphocyte numbers/function and robustness of the immune response will be described through descriptive analysis of relationships between pre-defined variables.
Time Frame: ALC at baseline and vaccine response at least 21 days after last dose of vaccine
Population: 30 participants did not have ALC data collected at baseline evaluation because they had complete blood count (CBC) ordered without differential count.
Measure: Number; unit: percentagae of participants
Groups:
- ALC <1000 Cells/mm³: Participants whose ALC was <1000 cells/mm³ were analyzed.
- ALC ≥1000 Cells/mm³: Participants whose ALC was ≥1000 cells/mm³ were analyzed.
Arm/Group | ALC <1000 Cells/mm³ | ALC ≥1000 Cells/mm³
Number analyzed (Participants) | 26 | 28
percentagae of participants | 62 | 68
Statistical Analysis 1: Comparison: ALC <1000 Cells/mm³ vs ALC ≥1000 Cells/mm³; Test type: Superiority or Other; p = 0.78, Fisher Exact

6. Primary Outcome: Rate of Seroprotection After 1 Dose of Vaccine
Description: The immune response of Fluzone HD to Fluzone was determined using the hemagglutination-inhibition (HAI) assay to each of the 3 antigens contained in the vaccine: H1, H3 and B. Seroprotection was defined as a post-vaccine HAI titer ≥40.
Time Frame: at least 21 days after first dose, which is given at the time of baseline evaluation visit, and prior to second dose
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Leukemia-HD | Leukemia-SD | Solid Tumor-HD | Solid Tumor-SD | HIV-HD | HIV-SD
Number analyzed (Participants) | 13 | 13 | 8 | 9 | 18 | 20
Percentage of participants
  H1 antigen | 77 | 85 | 75 | 78 | 100 | 100
  H3 antigen | 92 | 92 | 75 | 89 | 100 | 100
  B antigen | 62 | 85 | 63 | 89 | 100 | 90

7. Primary Outcome: Number of Participants Achieving Seroprotection After Second Dose of Vaccine
Description: as for outcome 6
Time Frame: 21 to 42 days after second dose
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | Leukemia-HD | Leukemia-SD | Solid Tumor-HD | Solid Tumor-SD | HIV-HD | HIV-SD
Number analyzed (Participants) | 13 | 13 | 8 | 9 | 18 | 20
number of participants
  H1 antigen | 11 | 12 | 7 | 9 | 18 | 19
  H3 antigen | 8 | 8 | 7 | 7 | 18 | 19
  B antigen | 10 | 10 | 6 | 8 | 18 | 19

8. Secondary Outcome: Rate of Vaccine Response by Seroprotection Compared by Absolute Lymphocyte Count (ALC)
Description: as for outcome 5
Time Frame: ALC at baseline and vaccine response at least 21 days after last dose of vaccine
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | ALC <1000 Cells/mm³ | ALC ≥1000 Cells/mm³
Number analyzed (Participants) | 26 | 28
percentage of participants | 96 | 100
Statistical Analysis 1: Comparison: ALC <1000 Cells/mm³ vs ALC ≥1000 Cells/mm³; Test type: Superiority or Other; p = 0.48, Fisher Exact

9. Secondary Outcome: Number of Local Reactogenicity Events After First Dose
Description: Number of moderate or greater local reactogenicity events associated with the administration of Fluzone or FluzoneHD. Local reactions were defined as pain, redness, or induration.
Time Frame: First 14 days after vaccination
Measure: Number; unit: Events
Arm/Group | High-dose FluzoneHD | Standard Dose Fluzone
Number analyzed (Participants) | 41 | 42
Events | 19 | 16
Statistical Analysis 1: Comparison: High-dose FluzoneHD vs Standard Dose Fluzone; Test type: Superiority or Other; p = 0.51, Fisher Exact

10. Secondary Outcome: Number of Local Reactogenicity Events After Second Dose
Description: as for outcome 9
Time Frame: First 14 days after vaccination
Measure: Number; unit: Events
Arm/Group | High-dose FluzoneHD | Standard Dose Fluzone
Number analyzed (Participants) | 39 | 40
Events | 11 | 7
Statistical Analysis 1: Comparison: High-dose FluzoneHD vs Standard Dose Fluzone; Test type: Superiority or Other; p = 0.29, Fisher Exact

11. Secondary Outcome: Number of Systemic Reactogenicity Events After First Dose
Description: Number of moderate or greater systemic reactogenicity event associated with the administration of Fluzone or FluzoneHD. Systemic reactions were defined as muscle ache, fatigue, or fever.
Time Frame: First 14 days after vaccination
Measure: Number; unit: Events
Arm/Group | High-dose FluzoneHD | Standard Dose Fluzone
Number analyzed (Participants) | 41 | 42
Events | 10 | 7
Statistical Analysis 1: Comparison: High-dose FluzoneHD vs Standard Dose Fluzone; Test type: Superiority or Other; p = 0.43, Fisher Exact

12. Secondary Outcome: Number of Systemic Reactogenicity Events After Second Dose
Description: as for outcome 11
Time Frame: First 14 days after vaccination
Measure: Number; unit: Events
Arm/Group | High-dose FluzoneHD | Standard Dose Fluzone
Number analyzed (Participants) | 39 | 40
Events | 8 | 3
Statistical Analysis 1: Comparison: High-dose FluzoneHD vs Standard Dose Fluzone; Test type: Superiority or Other; p = 0.11, Fisher Exact

13. Secondary Outcome: Comparison of Geometric Mean Titer (GMT) by HAI
Description: Serum antibody levels expressed as the reciprocal of the dilution needed to inhibit hemagglutination in vitro.
Time Frame: Pre-vaccination, post-vaccination and 9 months after vaccination
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Titers
Groups:
- Solid Tumor-HD; Solid Tumor-SD: Patients with a diagnosis of solid tumor who received the standard dose Fluzone.
Arm/Group | Leukemia-HD | Leukemia-SD | Solid Tumor-HD | Solid Tumor-SD | HIV-HD | HIV-SD
Number analyzed (Participants) | 13 | 13 | 8 | 9 | 18 | 20
Titers
  H1 Antigen/Pre-vaccination | 29 [17 to 49] | 50 [22 to 111] | 57 [16 to 203] | 40 [20 to 81] | 71 [37 to 137] | 67 [40 to 113]
  H1 Antigen/Post-vaccination | 117 [62 to 221] | 161 [82 to 317] | 580 [157 to 2137] | 148 [84 to 260] | 373 [264 to 528] | 267 [188 to 378]
  H1 Antigen/9 Months Post-vaccination | 30 [11 to 87] | 85 [14 to 533] | 403 [33 to 4940] | 80 [12 to 533] | 279 [145 to 535] | 174 [93 to 325]
  H3 Antigen/Pre-vaccination | 26 [12 to 58] | 25 [10 to 61] | 20 [6 to 69] | 22 [9 to 53] | 42 [24 to 72] | 49 [31 to 78]
  H3 Antigen/Post-vaccination | 139 [49 to 394] | 63 [21 to 188] | 215 [104 to 445] | 109 [31 to 381] | 154 [105 to 226] | 143 [97 to 212]
  H3 Antigen/9 Months Post-vaccination | 49 [16 to 148] | 40 [13 to 123] | 101 [28 to 360] | 143 [49 to 416] | 70 [44 to 111] | 102 [52 to 199]
  B Antigen/Pre-vaccination | 16 [8 to 31] | 29 [15 to 57] | 17 [8 to 35] | 23 [12 to 47] | 33 [23 to 48] | 34 [23 to 48]
  B Antigen/Post-vaccination | 181 [89 to 371] | 113 [36 to 357] | 195 [33 to 1138] | 202 [83 to 488] | 160 [108 to 237] | 172 [100 to 297]
  B Antigen/9 Months Post-vaccination | 9 [6 to 13] | 13 [6 to 28] | 16 [6 to 43] | 11 [5 to 23] | 13 [9 to 19] | 13 [9 to 19]

14. Secondary Outcome: Comparison of Geometric Mean Ratios (GMR) by HAI
Description: GMTs compared to each other as a ratio of the pre- and post-vaccine titers and as the ratio post-last dose to 9 months later.
  GMRs were compared pre- to post-vaccination and post- vaccination to 9 months later.
Time Frame: Pre-vaccination, post-vaccination and 9 months after vaccination
Population: as for outcome 1
Measure: Number; unit: Ratio
Arm/Group | Leukemia-HD | Leukemia-SD | Solid Tumor-HD | Solid Tumor-SD | HIV-HD | HIV-SD
Number analyzed (Participants) | 13 | 13 | 8 | 9 | 18 | 20
Ratio
  H1 post- over pre-vaccination | 4.0 | 3.2 | 10.2 | 3.7 | 5.2 | 4.0
  H1 post-vaccination over 9 months | 3.9 | 1.9 | 1.4 | 1.9 | 1.3 | 1.5
  H3 post- over pre-vaccination | 5.3 | 2.6 | 10.8 | 5.0 | 3.7 | 2.9
  H3 post-vaccination over 9 months | 2.8 | 1.6 | 2.1 | 0.8 | 2.2 | 1.4
  B post- over pre-vaccination | 11.2 | 3.9 | 11.6 | 8.6 | 4.8 | 5.1
  B post-vaccination over 9 months | 20.6 | 8.8 | 12.3 | 18.0 | 12.1 | 12.9

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 21 days after each dose of vaccine. No "other" adverse events were observed.
Arm/Group | Leukemia-HD | Leukemia-SD | Solid Tumor-HD | Solid Tumor-SD | HIV-HD | HIV-SD
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 1/8 | 0/9 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/8 | 0/9 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leukemia-HD (N=13) | Leukemia-SD (N=13) | Solid Tumor-HD (N=8) | Solid Tumor-SD (N=9) | HIV-HD (N=20) | HIV-SD (N=20)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — In 9-year-old with history of neurologic disorder who received FluzoneHD after recovery from sedation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes